CLINICAL TRIAL: NCT00726141
Title: Brief Interventions on Smoking for Hormonal Contraceptive Users
Acronym: BRISC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Luebeck (Other)
Responsible Party: PD Dr. Hans-Jürgen Rumpf, University of Lübeck, Research group S:TEP (Substance misuse: Treatment, Epidemiology and Prevention)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 01EB0421; BMBF grant no: 01EB0421
Record Dates: First submitted 2008-07-28; First posted 2008-07-31 (Estimated); Last update posted 2008-07-31 (Estimated); Status verified 2008-07

CONDITIONS: Smoking
Keywords: Brief Intervention; Smoking Cessation; Motivational Interviewing; Expert System; Readiness to Change; Hormonal Contraceptive; Adolescents
MeSH Terms: conditions — Smoking; Smoking Cessation | interventions — Crisis Intervention; Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Brief intervention, Motivational Interviewing, Expert System — Motivational Interviewing, stage-tailored self-help manual, physician letter, expert system feedback letter

SUMMARY:
Despite rising smoker rates, particularly in girls and young women, only few studies have focused on smoking cessation in young smokers. Gynaecologist practices may be an ideal setting to proactively intervene with young female smokers. Elevated health risks of smoking while using hormonal contraceptives could be a successful approach to gain young women's attention on smoking cessation. The purpose of this study is to evaluate the effectiveness of a smoking cessation intervention for girls and young women visiting gynaecologist practices and using hormonal contraceptives.

DETAILED DESCRIPTION:
In the randomized controlled trial, female smokers aged 14-25 will be recruited in practices of gynaecologists. Intervention within the practice consists of a 30 minutes counseling session based on Motivational Interviewing, a standardised physician letter focusing on the elevated health risks of smoking while using hormonal contraceptives and a stage-matched self-help manual. After four weeks, an expert system feedback letter will be sent. In the intervention group, no smoking intervention will be given. Follow-up assessments will be conducted after 12 months, including saliva cotinine measures.

ELIGIBILITY:
Inclusion Criteria

* Age 14-25
* Having smoked at least 1 cigarette within last 4 weeks
* Use of hormonal contraceptives or intention for prescription within next 2 weeks

Exclusion Criteria:

* Pregnancy
* Emergency treatment

Ages: 14 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 699 (Actual)
Dates: Start 2004-10; Primary Completion 2005-01 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Smoking cessation | 12 months

SECONDARY OUTCOMES:
Reduction of smoking | 12 months
Readiness to change variables | 12 months
Level of nicotine dependence | 12 months
Quit attempts | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: PD Dr. Hans-Jürgen Rumpf, Dipl.-Psych., Principal Investigator — University of Luebeck
Locations (1):
- University of Lübeck, Lübeck, Germany